CLINICAL TRIAL: NCT04166461
Title: Assessment of Esophageal Mucosal Impedance Before and After Sleeve Gastrectomy
Brief Title: Mucosal Impedance Sleeve Gastrectomy
Status: Recruiting | Type: Observational
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, RONNIE FASS, Professor of Medicine, Gastroenterology Department Chair, MetroHealth Medical Center
Other Study IDs: IRB19-00589
Record Dates: First submitted 2019-11-14; First posted 2019-11-18 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Gastroesophageal Reflux; Bariatric Surgery Candidate
Keywords: Mucosal impedance; Sleeve gastrectomy; GERD
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Not application, observational study — Not application, observational study

SUMMARY:
Obesity is a growing epidemic and bariatric surgery has been shown to be the most effective and efficient mean of achieving significant and sustainable weight loss in morbidly obese individuals. Studies have demonstrated that after LSG, between 5 and 30% of patients suffered from GERD, with a small subset of those patients (2.9 %) converting to another bariatric procedure (gastric bypass) because of debilitating GERD symptoms.

The investigators propose this current study to examine mucosal impedance before and after sleeve gastrectomy using the novel mucosal impedance procedure, as well as assess quality of life and GERD symptoms parameters. In addition, this study will determine if the level of mucosal impedance pre-sleeve gastrectomy may predict the development of GERD post-surgery. Our Hypothesis is that sleeve gastrectomy is highly associated with the risk of developing new onset GERD.

This is a prospective, comparative cohort study. A total of 15 obese patients (BMI ≥ 35) undergoing sleeve gastrectomy by choice will be recruited into the study from our bariatric and weight management program. An initial screening upper endoscopy will be performed as part of pre-bariatric evaluation, during which mucosal impedance will be performed with the consent of the patient. Patients with evidence of erosive esophagitis (LA grade A-D), Barrett's esophagus or eosinophilic esophagitis will be excluded from the study. As per surgical recommendation, PPI will be used for 6 months in all bariatric patients.

Six months post-surgery, study patients will be re-evaluated by the GERD symptoms Checklist and SF 36. In addition, their new BMI will be documented. PPI will be held for at least 1 week and a 6 months post-surgical upper endoscopy will be performed to determine the presence or absence of erosive esophagitis and Barrett's esophagus. In addition, esophageal mucosal impedance will be reassessed.

DETAILED DESCRIPTION:
Rationale/Significance:

Obesity is a growing epidemic problem around the world. World Health Organization (WHO) defines obesity as a body mass index (BMI) over 30 Kg/m2 and it is estimated that 10% of the world's population is obese. Associated with obesity are health conditions that carry significant morbidity and mortality, including cardiovascular disease, osteoarthritis, diabetes, cancer (breast, colon and endometrial) and gastroesophageal reflux disease (GERD). Bariatric surgery has been shown to be the most effective and efficient mean of achieving significant and sustainable weight loss in morbidly obese individuals.

As part of their limited GI workup, candidates for bariatric surgery usually undergo only an upper endoscopy prior to surgery. However, no studies are preferred to assess the degree of esophageal acid exposure in patients with normal endoscopy who are candidates for LSG. In addition, there is no routine assessment of patients post LSG for the development of GERD.

The effect of laparoscopic sleeve gastrectomy (LSG) on GERD has been equivocal with low-quality evidence suggesting both improvement and worsening of reflux after surgery. Studies have demonstrated that after LSG, between 5 and 30% of patients suffered from GERD, with a small subset of those patients (2.9 %) converting to another bariatric procedure (gastric bypass) because of debilitating GERD symptoms.

As part of their limited GI workup, candidates for bariatric surgery usually undergo only an upper endoscopy prior to surgery. Currently there is no routine formal (endoscopic or pH) assessment of patients after gastric weight loss surgery for the development of GERD. The effect of laparoscopic sleeve gastrectomy (LSG) on GERD has been equivocal with low-quality evidence from various studies suggesting both improvement and worsening of reflux after surgery.

The main purpose of this study is to evaluate whether GERD develops after LSG and to examine the esophagus after LSG for the possible development of acid reflux both endoscopically (visible by camera view) and on a cellular level by obtaining mucosal impedance. Mucosal impedance (MI) is a measurement that can evaluate if the structure of the esophageal tissue is normal or abnormal. MI is performed using an FDA approved endoscopic tool called "Mucosal Integrity Conductivity Test System" (Diversatek). The MI system software uses the collected data to determine if there is evidence of GERD.

Objective:

The investigators propose this current study to examine mucosal impedance before and after sleeve gastrectomy using the novel mucosal impedance procedure, as well as assess quality of life and GERD symptoms parameters. In addition, this study will determine if the level of mucosal impedance pre-sleeve gastrectomy may predict the development of GERD post-surgery. Our Hypothesis is that sleeve gastrectomy is highly associated with the risk of developing new onset GERD.

This is a prospective, comparative cohort study. A total of 15 obese patients (BMI ≥ 35) undergoing sleeve gastrectomy by choice will be recruited into the study from our bariatric and weight management program. An initial screening upper endoscopy will be performed as part of pre-bariatric evaluation, during which mucosal impedance will be performed with the consent of the patient. Patients with evidence of erosive esophagitis (LA grade A-D), Barrett's esophagus or eosinophilic esophagitis will be excluded from the study. As per surgical recommendation, PPI will be used for 6 months in all bariatric patients.

Six months post-surgery, study patients will be re-evaluated by the GERD symptoms Checklist and SF 36. In addition, their new BMI will be documented. PPI will be held for at least 1 week and a 6 months post-surgical upper endoscopy will be performed to determine the presence or absence of erosive esophagitis and Barrett's esophagus. In addition, esophageal mucosal impedance will be reassessed.

Primary aim

- To determine the development of GERD after sleeve gastrectomy by measuring esophageal mucosal impedance pre and post-surgery.

Secondary aim

* To determine the degree of GERD development post sleeve gastrectomy
* To determine any effect on quality of life post-sleeve gastrectomy

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory male or female (non-pregnant) and is 18-80 years old at the time of enrollment.
* Adults with BMI 35 ≥ kg/m2
* Patients scheduled for sleeve gastrectomy
* Patients with no presence of esophagitis on screening upper endoscopy will be recruited to pursue 6mo- post-op upper endoscopy.

Exclusion Criteria:

* Age < 18 or > 80 years old
* Female patients cannot be pregnant or agree to avoid pregnancy during study period.
* History of GERD, erosive esophagitis, esophageal stricture, Barrett's esophagus or esophageal varices
* History of a major motility disorder: achalasia, diffuse esophageal spasm, jackhammer esophagus, esophagogastric junction outflow obstruction, and absent peristalsis.
* History of Eosinophilic Esophagitis
* History of bariatric surgery or other upper gastrointestinal surgery
* History of Scleroderma
* PPI use prior to bariatric procedure
* History of severe psychiatric disorder, including suicidal ideation or admission to psychiatric institution.
* Negative upper endoscopy during pre-LSG evaluation for esophagitis, Barrett's esophagus, peptic stricture or eosinophilic esophagitis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include patients from the Metrohealth Medical Center bariatric and weight management program who are candidates for sleeve gastrectomy.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-04-21 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
Development of gastroesophageal reflux disease after sleeve gastrectomy | Time of recruitment to 6 months after sleeve gastrectomy
  On second esophagogastroduodenoscopy, visualized esophagitis would indicate development of gastroesophageal reflux disease.

SECONDARY OUTCOMES:
Level of GERD and quality of life after sleeve gastrectomy | Time of recruitment to 6 months after sleeve gastrectomy
  These measures would be obtained through surveys during follow up period.

CONTACTS AND LOCATIONS:
Overall Officials: Ronnie Fass, MD, Principal Investigator — MetroHealth Medical Center
Locations (1):
- MetroHealth - Main Campus Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No